CLINICAL TRIAL: NCT02002767
Title: A Phase 1, Open-Label, Parallel-Group, Single-Dose Study to Evaluate the Pharmacokinetics of GS-5816 in Subjects With Normal Renal Function and Severe Renal Impairment
Brief Title: Study to Evaluate the Pharmacokinetics of Velpatasvir in Participants With Normal Renal Function and Severe Renal Impairment
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Gilead Sciences (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GS-US-281-1056; 2013-004113-41 (EudraCT Number)
Record Dates: First submitted 2013-12-02; First posted 2013-12-06 (Estimated); Results first posted 2020-11-16 (Actual); Last update posted 2020-11-16 (Actual); Status verified 2020-10

CONDITIONS: Hepatitis C Virus
MeSH Terms: conditions — Hepatitis C | interventions — velpatasvir

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Participants with renal impairment (Experimental): Participants with severe renal impairment will receive a single dose of velpatasvir.
  Interventions: Drug: Velpatasvir
- Participants with normal renal function (Active Comparator): Participants with normal renal function will receive a single dose of velpatasvir.
  Interventions: Drug: Velpatasvir

INTERVENTIONS:
Drug: Velpatasvir — Velpatasvir 100 mg (2 x 50 mg tablets) administered orally
  Other Names: GS-5816

SUMMARY:
The primary objective of the study is to evaluate the single-dose pharmacokinetics (PK) of velpatasvir (formerly GS-5816) in participants with severe renal impairment using matched healthy participants as a control group.

ELIGIBILITY:
Key Inclusion Criteria:

* General good health with stable chronic kidney disease in Severe Renal Impairment Group
* Screening labs within defined thresholds
* Creatinine clearance must be < 30 mL/min for Severe Renal Impairment group, and ≥ 90 mL/min for Normal Renal Function group

Key Exclusion Criteria:

* Females who are pregnant or nursing, or males who have a pregnant partner
* Infection with hepatitis B virus (HBV), hepatitis C virus (HCV) or HIV
* History of clinically significant illness (including psychiatric or cardiac) or any other medical disorder that may interfere with participant treatment and/or adherence to the protocol

Note: Other protocol defined Inclusion/Exclusion criteria may apply.

Ages: 18 Years to 79 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2013-12-16 (Actual); Primary Completion 2014-06-09 (Actual); Study Completion 2014-06-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gilead Study Director, Study Director — Gilead Sciences
Locations (5):
- United States (4):
  - Miami, Florida
  - Orlando, Florida
  - Saint Paul, Minnesota
  - San Antonio, Texas
- Christchurch, New Zealand

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled at study sites in United Stated and New Zealand. The first participant was screened on 16 December 2013. The last study visit occurred on 09 June 2014.
Pre-assignment Details: 46 participants were screened.
Groups:
- Normal Renal Function: Participants with normal renal function received velpatasvir 100 mg administered orally with a light breakfast on Day 1.
- Severe Renal Impairment: Participants with severe renal impairment received velpatasvir 100 mg administered orally with a light breakfast on Day 1.
Period: Overall Study
Arm/Group | Normal Renal Function | Severe Renal Impairment
Started | 9 | 10
Completed | 9 | 10
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: The Safety Analysis Set included participants who were enrolled and received at least 1 dose of study drug.
Groups:
- Total: Total of all reporting groups
Arm/Group | Normal Renal Function | Severe Renal Impairment | Total
Number analyzed (Participants) | 9 | 10 | 19
Age, Continuous [Mean (Standard Deviation); unit: years] | 66 (3.7) | 71 (4.0) | 68 (4.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 5 | 10
  Male | 4 | 5 | 9
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Not Hispanic or Latino | 5 | 7 | 12
  Hispanic or Latino | 4 | 3 | 7
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Black or African American | 1 | 2 | 3
  White | 8 | 8 | 16

OUTCOME MEASURES:

1. Primary Outcome: Pharmacokinetic (PK) Parameter of Velpatasvir: AUClast
Description: AUClast is defined as the area under the plasma concentration versus time curve from time zero to the last quantifiable concentration.
Time Frame: Pre-dose (≤ 5 min), 0.5, 1, 2, 2.5, 3, 3.5, 4, 6, 8, 12, 18, 24, 48, 72, 96, and 120 hours post-dose on Day 1
Population: The PK analysis set included all enrolled and treated participants who have evaluable PK profiles for velpatasvir.
Measure: Mean (Standard Deviation); unit: h*ng/mL
Arm/Group | Normal Renal Function | Severe Renal Impairment
Number analyzed (Participants) | 9 | 10
h*ng/mL | 5597.8 (1749.18) | 7971.7 (2531.09)
Statistical Analysis 1: Comparison: Normal Renal Function vs Severe Renal Impairment; A sample size of 8 evaluable participants in each renal function group (normal and severely impaired) will provide at least 80% power to reject the null hypothesis that participants with severe renal impairment have a minimum increase of 100% in AUC0-last, AUCinf, or Cmax of velpatasvir compared to participants with normal renal function; Test type: Other; Geometric Least Squares Mean(GLSM) Ratio = 149.05, 90% CI 2-sided [116.62 to 190.49]

2. Primary Outcome: PK Parameter of Velpatasvir: AUCinf
Description: AUCinf is defined as the area under the plasma concentration versus time curve extrapolated to infinite time.
Time Frame: Pre-dose (≤ 5 min), 0.5, 1, 2, 2.5, 3, 3.5, 4, 6, 8, 12, 18, 24, 48, 72, 96, and 120 hours post-dose on Day 1
Population: Participants in the PK Analysis Set were analyzed.
Measure: Mean (Standard Deviation); unit: h*ng/mL
Arm/Group | Normal Renal Function | Severe Renal Impairment
Number analyzed (Participants) | 9 | 10
h*ng/mL | 5651.6 (1763.12) | 8108.3 (2628.18)
Statistical Analysis 1: Comparison: Normal Renal Function vs Severe Renal Impairment; [analysis description as in outcome 1, analysis 1]; Test type: Other; GLSM Ratio = 149.90, 90% CI 2-sided [116.97 to 192.11]

3. Primary Outcome: PK Parameter of Velpatasvir: Cmax
Description: Cmax is defined as the maximum observed plasma concentration of drug.
Time Frame: Pre-dose (≤ 5 min), 0.5, 1, 2, 2.5, 3, 3.5, 4, 6, 8, 12, 18, 24, 48, 72, 96, and 120 hours post-dose on Day 1
Population: Participants in the PK Analysis Set were analyzed.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Normal Renal Function | Severe Renal Impairment
Number analyzed (Participants) | 9 | 10
ng/mL | 702.7 (197.20) | 732.4 (176.19)
Statistical Analysis 1: Comparison: Normal Renal Function vs Severe Renal Impairment; [analysis description as in outcome 1, analysis 1]; Test type: Other; GLSM Ratio = 110.85, 90% CI 2-sided [90.76 to 135.38]

4. Secondary Outcome: Percentage of Participants Experiencing Treatment-Emergent Adverse Events
Description: Treatment-emergent adverse events (TEAEs) were defined as any adverse events (AEs) with an onset date on or after the study drug start date and no later than 30 days after permanent discontinuation of study drug.
Time Frame: First dose date plus 30 days
Population: The Safety Analysis Set included participants who were enrolled and received at least 1 dose of study drug.
Measure: Number; unit: percentage of participants
Arm/Group | Normal Renal Function | Severe Renal Impairment
Number analyzed (Participants) | 9 | 10
percentage of participants | 0 | 20

5. Secondary Outcome: Percentage of Participants Experiencing Treatment-Emergent Laboratory Abnormalities
Description: A treatment-emergent laboratory abnormality was defined as an increase of at least 1 abnormality grade from baseline and occurring after the first dose of study drug and within 30 days after last study drug administration. The severity of laboratory abnormalities was assessed as Grade 0, 1 (mild), 2 (moderate), 3 (severe), or 4 (potentially life threatening).
Time Frame: First dose date plus 30 days
Population: Participants in the Safety Analysis Set were analyzed.
Measure: Number; unit: percentage of participants
Arm/Group | Normal Renal Function | Severe Renal Impairment
Number analyzed (Participants) | 9 | 10
percentage of participants
  Grade 1 | 33.3 | 20
  Grade 2 | 0 | 30
  Grade 3 | 0 | 30
  Grade 4 | 0 | 10

6. Secondary Outcome: Percentage Protein Binding of Velpatasvir
Description: Mean velpatasvir protein binding (percentage free and percentage bound) was determined in all participants at 2 or 3 hours post-dose. Protein binding was assessed at Tmax whenever possible or at the time point closest to Tmax for each participant.
Time Frame: 2 or 3 hours post-dose on Day 1
Population: Participants in the PK Analysis Set were analyzed.
Measure: Mean (Standard Deviation); unit: percentage of plasma protein binding
Arm/Group | Normal Renal Function | Severe Renal Impairment
Number analyzed (Participants) | 9 | 10
percentage of plasma protein binding
  Free Protein Percentage | 0.29 (0.012) | 0.29 (0.012)
  Bound Protein Percentage | 99.71 (0.012) | 99.71 (0.012)

ADVERSE EVENTS:
Time Frame: First dose date plus 30 days
Description: The Safety Analysis Set included participants who were enrolled and received at least 1 dose of study drug.
Arm/Group | Normal Renal Function | Severe Renal Impairment
All-Cause Mortality (participants affected / at risk) | 0/9 | 0/10
Serious Adverse Events (participants affected / at risk) | 0/9 | 0/10
Other Adverse Events (participants affected / at risk) | 0/9 | 2/10
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Normal Renal Function (N=9) | Severe Renal Impairment (N=10)
Vessel puncture site haemorrhage (General disorders) | 0 | 1
Dizziness (Nervous system disorders) | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
After conclusion of the study and without prior written approval from Gilead, investigators in this study may communicate, orally present, or publish in scientific journals or other media only after the following conditions have been met:

* The results of the study in their entirety have been publicly disclosed by or with the consent of Gilead in an abstract, manuscript, or presentation form; or
* The study has been completed at all study sites for at least 2 years